CLINICAL TRIAL: NCT00537654
Title: An Open-Label, Randomized, Single Dose Three-Period Partial Crossover Study to Determine the Bioequivalence and Food Effect of a Combination Capsule Formulation of Dutasteride and Tamsulosin Hydrochloride (0.5mg/0.4mg) Compared to Concomitant Dosing of AVODART™ 0.5mg and Flomax 0.4mg Commercial Capsules in Healthy Male Subjects
Brief Title: A Study To Compare Giving AVODART And FLOMAX Together Or In A Combination Capsule In The Fed And Fasted State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARI109882
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia,; AVODART,; FLOMAX
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted state (Experimental): Subjects will be required to fast overnight. Subjects will participate in 3 treatment periods and assigned to one of 12 treatment sequences ( ABC, ACB, BAC, BCA, CAB, CBA, ABD, ADB, BAD, BDA, DAB, DBA) in accordance with the randomization schedule. The three treatment periods will be separated by a minimum washout period of 28 days
  Interventions: Drug: Treatment sequence C; Drug: Treatment sequence D
- Fed state (Experimental): Subjects will be served high fat breakfast 30 minutes prior to dosing. Subjects will participate in 3 treatment periods and assigned to one of 12 treatment sequences ( ABC, ACB, BAC, BCA, CAB, CBA, ABD, ADB, BAD, BDA, DAB, DBA) in accordance with the randomization schedule. The three treatment periods will be separated by a minimum washout period of 28 days
  Interventions: Drug: Treatment sequence A; Drug: Treatment sequence B

INTERVENTIONS:
Drug: Treatment sequence A — Commercially available tamsulosin hydrochloride 0.4 mg and dutasteride 0.5 mg in a fed state
  Arms: Fed state
Drug: Treatment sequence B — Fixed dose combination formulation of dutasteride and tamsulosin hydrochloride (0.5 mg dutasteride, 0.4 mg tamsulosin hydrochloride) in a fed state
  Arms: Fed state
Drug: Treatment sequence C — Commercially available tamsulosin hydrochloride 0.4 mg and dutasteride 0.5 mg in a fasted state
  Arms: Fasted state
Drug: Treatment sequence D — Fixed dose combination formulation of dutasteride and tamsulosin hydrochloride (0.5 mg dutasteride, 0.4 mg tamsulosin hydrochloride) in a fasted state
  Arms: Fasted state

SUMMARY:
This study will be an open-label, randomized, single dose, three way partial crossover study in healthy male subjects. The aim of the study is to evaluate bioequivalence of a fixed dose combination (FDC) capsule of dutasteride and tamsulosin hydrochloride (HCl) (0.5 milligram [mg]/0.4 mg) relative to co-administration of dutasteride 0.5 mg capsules and tamsulosin hydrochloride 0.4 mg tablets in both the fed and fasted states. Approximately 98 healthy adult male subjects will be enrolled into the study. Subjects will receive single oral doses in 3 treatment periods and be randomized to one of twelve different treatment sequences (ABC, ACB, BAC, BCA, CAB, CBA, ABD, ADB, BAD, BDA, DAB, DBA) wherein A= commercially available tamsulosin hydrochloride 0.4 mg and dutasteride 0.5 mg in a fed state, B= fixed dose combination formulation of dutasteride and tamsulosin hydrochloride (0.5 mg dutasteride, 0.4 mg tamsulosin hydrochloride) in a fed state, C= commercially available tamsulosin hydrochloride 0.4 mg and dutasteride 0.5 mg in a fasted state, D= fixed dose combination formulation of dutasteride and tamsulosin hydrochloride (0.5 mg dutasteride, 0.4 mg tamsulosin hydrochloride) in a fasted state. Each treatment period will be separated by a minimum 28 day washout period. The total duration of a subject's involvement in this study is approximately 15-18 weeks.

DETAILED DESCRIPTION:
An Open-Label, Randomized, Single Dose Three-Period Partial Crossover Study to Determine the Bioequivalence and Food Effect of a Combination Capsule Formulation of Dutasteride and Tamsulosin Hydrochloride (0.5mg/0.4mg) Compared to Concomitant Dosing of AVODART 0.5mg and FLOMAX 0.4mg Commercial Capsules in Healthy Male Subjects

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects defined as individuals who are free from clinically significant illness or disease as determined by the investigator based on their medical history, physical examination, laboratory studies, ECGs, and other tests.
* Males who are 18 - 45 years of age, inclusive.
* Weight range 55 - 95 kg (inclusive) and body mass index 19 - 30 kg/m2 (inclusive).
* Willing and able to give written informed consent, willing to participate for the full duration of the study, and able to understand and follow instructions related to study procedures

Exclusion criteria:

* Slow metabolizer for CYP2D6 as determined by screening PGx analysis.
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer, such as St. John's Wort) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Chronic hepatitis B and C, as evidence by positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody.
* Positive HIV test at screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of regular alcohol consumption exceeding 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening. Subjects must be able and willing to abstain from beverages and foods containing alcohol 24 hours prior to and during the dosing day.
* A positive urine drug or alcohol (Breath test or urine) screen result at screening or check-in..
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication or anytime during the study period.
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.
* History or presence of allergy, intolerance, or contraindication to tamsulosin HCl or AVODART or drugs of this class, or a history of drug or other allergy (including true sulfonamide allergy) that, in the opinion of the physician responsible, contraindicates their participation.
* Subjects who have consumed the following foods or drinks within 7 days prior to the first dose of study medication or at any time during the clinical phase of the study: grapefruit juice; red wine; grapefruit or cruciferous vegetables (watercress, broccoli, cabbage, Brussels sprouts).
* QTc ≥ 450 msec at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2007-10-18 (Actual); Primary Completion 2008-02-22 (Actual); Study Completion 2008-02-22 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) from time zero to 24 hours (AUC[0-24]) of plasma tamsulosin in fed state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Area under the curve from time zero to infinity (AUC[0-inf]) of plasma tamsulosin in fed state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Concentration maximum (Cmax) of plasma tamsulosin in fed state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Area under the curve (AUC) from time zero to 24 hours (AUC[0-24]) of plasma dutasteride in fed state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Area under the curve (AUC) from time zero to 72 hours (AUC[0-72]) of plasma dutasteride in fed state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Concentration maximum (Cmax) of plasma dutasteride in fed state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Area under the curve (AUC) from time zero to 24 hours (AUC[0-24]) of plasma tamsulosin in fasted state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Area under the curve from time zero to infinity (AUC[0-inf]) of plasma tamsulosin in fasted state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Concentration maximum (Cmax) of plasma tamsulosin in fasted state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Area under the curve (AUC) from time zero to 24 hours (AUC[0-24]) of plasma dutasteride in fasted state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Area under the curve (AUC) from time zero to 72 hours (AUC[0-72]) of plasma dutasteride in fasted state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Concentration maximum (Cmax) of plasma dutasteride in fasted state | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points

SECONDARY OUTCOMES:
Concentration minimum (Cmax) of plasma tamsulosin | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Time to maximum observed plasma drug concentration (tmax) of tamsulosin and dutasteride | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Elimination half-life (t1/2) of tamsulosin and dutasteride | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Negative slope of the terminal phase of tamsulosin and dutasteride | Pre-dose and post dose at 1,2,3,4,5,6,7,8,10,12,16,24,36,48,72hrs
  Plasma samples will be collected at indicated time points
Number of subjects with adverse event (AE) and serious adverse event (SAE). | Up to 18 weeks
  AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE.
Number of subjects with abnormal clinical laboratory parameters | Up to 18 weeks
  Blood samples will be collected to analyze aspartate aminotransferase (AST), alkaline Phosphatase (ALP), alanine aminotransferase (ALT), creatinine, blood urea nitrogen, creatine kinase, total bilirubin, direct bilirubin, total protein, albumin, glucose, sodium, potassium, calcium
Number of subjects with abnormal hematology laboratory parameters | Up to 18 weeks
  Blood samples will be collected to analyze White Blood Cells (WBC), neutrophils, basophils, eosionophils, lymphocytes, monocytes, Red Blood Cells (RBC) count, RBC indices, Day -1average red blood cell size (MCV), hemoglobin amount per red blood cell (MCH) hemoglobin, hematocrit, and platelet count
Number of subjects with abnormal urinalysis | Up to 18 weeks
  Urine samples will be collected to analyze specific gravity, pH, glucose, protein, blood and ketones
Blood pressure assessment as a measure of safety | Up to 18 weeks
  Systolic and diastolic blood pressure will be measured in a supine position at pre-dose, Days 2, 3, 4,5,6,7,43 and 85 post-dose
Measurement of pulse rate as a measure of safety | Up to 18 weeks
  Pulse rate will be measured in a supine position at pre-dose, Days 2, 3, 4,5,6,7,43 and 85 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study ARI109882 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/ARI109882?search=study&study_ids=ARI109882#rs
- Available data/document: Dataset Specification: ARI109882 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ARI109882 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ARI109882 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ARI109882 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ARI109882 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ARI109882 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ARI109882 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register